CLINICAL TRIAL: NCT02902354
Title: Changes in Central Arterial Pressure of Normotensive Women Taking Nifedipine for Tocolysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, MD, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 27468
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Tocolysis With Nifedipine
MeSH Terms: interventions — Nifedipine; Tocolysis; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nifedipine for tocolysis (Other): Only women receiving nifedipine (as standard of care) for tocolysis
  Interventions: Other: Nifedipine for tocolysis

INTERVENTIONS:
Other: Nifedipine for tocolysis — observational
  Other Names: Standard of care

SUMMARY:
To determine the central blood pressure changes in normotensive women who are receiving nifedipine for uterine contraction suppression

DETAILED DESCRIPTION:
Only women whom have been prescribed nifedipine tocolysis by their covering obstetrician will be approached to participate in the study.

The patient will take their nifedipine as scheduled, we will attain central arterial pressure reading in addition to arterial waveform measurements. These will be collected:

Before administration of the medication Every 20 minutes for 3 hours (total of 10 measurements)

-This timing will allow measurements through approximately 2 half lives Routine sphygmomanometry will also be completed at the testing times All of these measurements will be collected for study purposes, although the nurses will have the opportunity to record the routine blood pressure measurements for their charting/vital signs assessment if they desire.

Once the patient has been monitored for 3 hours, her participation in the study is considered complete and no additional information will be collected. Each patient will serve as her own control (blood pressure prior to administration of medication), no randomization will occur.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Currently receiving tocolysis with nifedipine (10 or 20mg q4-6 hours)

Exclusion Criteria:

* Multiple pregnancy
* Diagnosis of hypertensive disorder in pregnancy or blood pressures 140/90 or higher on -more than 2 occasions.
* Currently on antihypertensive medications (Nifedipine XL, labetalol, hydralazine, methyl-dopa, etc)
* Currently on other tocolytic medications (exp: magnesium, Indocin)
* Narcotic use
* Renal diseaseI
* Irregular heart rhythms or arrhythmias
* Peripheral arterial disease, leg artery disease
* Reynaud's phenomena
* Intense cold/hypothermia
* If there is a wound at location of where central arterial cuff would be placed or tonometer for carotid assessment
* Severe tachycardia (>120)
* Greater than 1st degree heart block
* Severe asthma
* Congestive heart failure or heart disease
* Lupus, rheumatoid arthritis
* Inability to adequately monitor BP
* Magnesium treatment

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To determine the central blood pressure changes in normotensive women who are receiving nifedipine for tocolysis. | every 20 min for 3 hours
  To determine the central blood pressure changes in normotensive women who are receiving nifedipine for tocolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No